CLINICAL TRIAL: NCT02076737
Title: Model-based Iterative Reconstruction (MB-IR VEOTM) in Ultra Low-dose Abdominal CT Versus Adaptative Statistical Iterative Reconstruction (ASIR): A Prospective Study for Acute Renal Colic
Acronym: VEOLITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0183; 2012-A01699-34
Record Dates: First submitted 2014-02-21; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Model-based Iterative Reconstruction (MB-IR VEOTM)
Keywords: Model-based iterative reconstruction MB-IR; VEOTM; Ultra low-dose; Abdominal CT; Dose reduction; Adaptative statistical iterative reconstruction ASIR; Acute renal colic
MeSH Terms: conditions — Renal Colic

ARMS (1):
- VEO (Experimental)
  Interventions: Device: Model-based iterative reconstruction (MB-IR VEOTM) on CT Discovery 750HD (GE Healthcare, Milwaukee, WI)

INTERVENTIONS:
Device: Model-based iterative reconstruction (MB-IR VEOTM) on CT Discovery 750HD (GE Healthcare, Milwaukee, WI)

SUMMARY:
The purpose of this study is to determine if Model-based iterative reconstruction (MB-IR VEOTM) in ultra low-dose abdominal CT as the same accuracy for the diagnosis of acute renal colic versus standard CT with adaptative statistical iterative reconstruction (ASIR).

DETAILED DESCRIPTION:
Renal colic is a common recurrent pathology in young patients, multi explored by imaging such as CT and abdominal radiography.

Abdominal MDCT(MultiDetector Computed Tomography) without injection is the gold standard in diagnosis of acute flank pain suspect of renal colic due to high sensitivity (96%) and excellent specificity (100%).

The increased use of medical imaging examinations using ionizing radiation (+57 % between 2002 and 2007) makes it essential to optimize protocols, including CT-scans which represents 10.1 % of procedures and 58 % of the collective effective dose.

Model-based iterative reconstruction (MB-IR VEOTM) (GE Healthcare, Milwaukee, WI) can use a low dose acquisition, reducing the effective dose delivered to the patient almost 80% comparing a standard CT with the last algorithm: adaptative statistical iterative reconstruction (ASIR).

MB-IR VEOTM shows great potential for substantially reducing radiation doses at routine abdominal CT. ASIR is limited in this regard owing to reduced image quality and diagnostic capability. Further investigation is needed to determine the optimal dose level for MBIR(Model Base Iterative Reconstruction) that maintains adequate diagnostic performance. In general, objective and subjective image quality measurements do not necessarily correlate with diagnostic performance at ultralow-dose CT.

Objective:

Prospective clinical study, equivalence between two CT protocols for the diagnosis of acute renal colic.

Show that a low dose acquisition with model based iterative reconstruction (MB-IR VeoTM) is as good as a standard CT with adaptative statistical iterative reconstruction (ASIR) in the diagnosis acute renal colic

ELIGIBILITY:
Inclusion Criteria:

* Informed and a written consent
* Acute flank pain needed abdominal CT exploration.

Exclusion Criteria:

* Juvenile patients
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
acute renal colic | at day 1

SECONDARY OUTCOMES:
Measure of dose-length product | at day 1
Measurements of subjective image quality | at day 1
Evaluation of visceral fat | at ady 1

CONTACTS AND LOCATIONS:
Overall Officials: Louis BOYER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France